CLINICAL TRIAL: NCT02353104
Title: The Effects of the Onion-Pumpkin Extract on Blood Pressure: An Open-label, Adaptive-design, Pilot Study
Brief Title: The Effects of the Onion-Pumpkin Extract on Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicus Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HORN1000
Record Dates: First submitted 2015-01-20; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Onion-Pumpkin Extract (Experimental): Take two capsules, twice daily before breakfast and dinner
  Interventions: Dietary Supplement: Onion-Pumpkin Extract

INTERVENTIONS:
Dietary Supplement: Onion-Pumpkin Extract

SUMMARY:
This open-label, adaptive-design, pilot study was designed to evaluate the effect of Onion-Pumpkin Extract in supporting healthy blood pressure as assessed by the change in systolic and diastolic blood pressures. The effect of the product on glucose metabolism, lipid levels, and antioxidant levels would also be determined. Tolerability and safety of the study product would also be investigated.

DETAILED DESCRIPTION:
Hypertension has become one of the most common diseases in the world and considered a public health challenge due to its association with morbidity and mortality and increased cost to society. Hypertension is the most important risk factor for cardiovascular diseases such as coronary heart disease, stroke, congestive heart failure, and peripheral vascular disease. One fourth of adults in the United States have high blood pressure and among these, the blacks and the elderly have higher incidence of hypertension. This condition is characterized by abnormally high blood pressure with the systolic greater than 140 mmHg and diastolic greater than 90 mmHg (1).

Lowering blood pressure has been linked to 35% to 40% reductions in the incidence of stroke, 20%-25% in myocardial infarction, and 50% in heart failure. Management of hypertension includes lifestyle modifications and pharmacological therapy and antihypertensive drugs. Lifestyle modifications such as weight reduction in overweight and obese individuals, 8-week diet of fruits, vegetables, low-fat dairy products, whole grain, poultry fish and nuts with limited fats, red meat and sweets, reduction in dietary sodium, physical activity, and moderation of alcohol consumption have been shown to lower blood pressure. There are several classes of antihypertensive drugs, including angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs) β-blockers (BBs), calcium channel blockers (CCBs) and the thiazide-class diuretics. Among these, the diuretic based therapy was more effective than other treatments in preventing cardiovascular diseases as demonstrated by the Antihypertensive and Lipid-lowering Treatment to prevent Heart Attack (ALLHAT) trial (1, 2).

Blood pressure can be lowered without using prescription drugs. Nutraceuticals have found their application in the treatment of hypertension. Omega-3 polyunsaturated fatty acids, omega-9 fatty acids, garlic, seaweed, and various vitamins and minerals have been shown to reduce blood pressure significantly (3).

Animal studies have demonstrated the potential benefits of onion in hypertensive rats. In one study involving rats fed with a control diet or a high-fat high-sucrose diet with or without Welsh onion for 4 weeks, lower blood pressure was observed in rats with onion diet, especially the green-leafy type. In addition, these rats have higher levels of nitric oxide (NO) metabolites in the urine and plasma, lower activity of NADH/NADPH oxidase in the aorta, and suppressed angiotensin II production (4). The mechanism of the antihypertensive effect of onion probably involves increased saving of NO (4, 5). A randomized, placebo-controlled, double-blind trial also demonstrated significant decrease in arterial blood pressure and reduction in plasma viscosity five hours after administration of a formulation containing onion and olive oil (6).

Pumpkin has been used as a traditional medicine and it is known for its antidiabetic, antitumor, antibacterial, anti-inflammatory, and antihypertensive properties (7). Animal studies confirmed that pumpkin seed oil supplementation resulted in lower systolic and diastolic blood pressure as well as improvements in lipid profile in both non-ovariectomized and ovariectomized rats (8). Using enzyme assays, it was demonstrated that pumpkin have moderate to high alpha-glucosidase and ACE inhibitory activities (9). A recent clinical trial involved postmenopausal women and the effects of supplemented pumpkin seed oil in cholesterol levels. The results of this trial showed that 12-week administration of 2g/day pumpkin seed oil led to a significant increase in HDL cholesterol and significant decrease in diastolic blood pressure. Pumpkin seed oil also improved menopausal symptom scores by decreasing hot flushes, headaches, and joint pains (10).

This open-label, adaptive-design, pilot study was designed to evaluate the effect of Onion-Pumpkin Extract in supporting healthy blood pressure as assessed by the change in systolic and diastolic blood pressures. The effect of the product on glucose metabolism, lipid levels, and antioxidant levels would also be determined. Tolerability and safety of the study product would also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 and ≤ 35 kg/m2
* Blood pressure:

  * SBP: 140-160 mmHg
  * DBP: 80-90 mmHg
* Judged by the Investigator to be in general good health on the basis of medical history
* Females of child bearing potential must agree to use appropriate birth control methods during the entire study period.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Subjects currently taking any antihypertensive medications
* Subjects taking prescription blood pressure, cholesterol and/or diabetes medication.
* Subjects currently taking dietary supplements or over the counter medication. (2 week washout allowed)
* History or presence of cancer in the prior two years.
* Recent history of (within 12 months) or strong potential for alcohol or substance abuse.
* Current tobacco smokers
* Participation in a clinical study with exposure to any non-registered drug product within 30 days prior.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk

  * Including subjects who are Bed or wheelchair-bound
* Clinically significant abnormal Physical Examination.
* Central Neurological disorders including but not limited to Spinal cord injuries, multiple sclerosis, and Parkinson disease.
* Pregnant, lactating, or unwilling to use adequate contraception during the duration of the study.
* Any other condition that, in the opinion of the investigator, would adversely affect the subject's ability to complete the study or its measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 12 weeks
  Change in Individual SBP Values
Systolic Blood Pressure (Change in Mean SBP Values) | 12 weeks
  Change in Mean SBP Values
Diastolic Blood Pressure (Change in Individual DBP Values) | 12 weeks
  Change in Individual DBP Values
Diastolic Blood Pressure (Change in Mean DBP Values) | 12 weeks
  Change in Mean DBP Values

SECONDARY OUTCOMES:
Change in complete blood cell count (CBC) | 12 weeks
Change in Comprehensive Metabolic Panel (CMP) | 12 weeks